CLINICAL TRIAL: NCT00667316
Title: Study to Identify the Influence of Different Factors on Workers' Disability Due to Low Back Pain
Brief Title: The Influence of Different Factors on Workers' Disability Due to Low Back Pain
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK-I-25
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
Keywords: low back pain; workers; disability; sick leave
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Workers from companies and workers' health care organizations who go for their periodic medical checkup.
  Interventions: Behavioral: Set of questionnaires (respondent)

INTERVENTIONS:
Behavioral: Set of questionnaires (respondent) — A set of questionnaires to determine risk factors for sick leave due to low back pain.

SUMMARY:
The purpose of this study is to determine, in Spanish workers, the influence of different factors (personal, psychological, work related and clinical) on the risk of being on sick leave during the 18 months after baseline assessment, and on the duration of that sick leave.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who get their checkups at participating health services
* With a labor contract that won't make it likely that they stop work before the next 18 months, for causes other than their health
* Who sign the informed consent form

Exclusion Criteria:

* Don't sign the informed consent form
* Inability to fill our the questionnaires
* Bedridden
* Rheumatologic inflammatory disease, cancer or fibromyalgia
* Suspicion of fibromyalgia
* Red flags for systemic disease
* Criteria for surgery
* Criteria for urgent referral to surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers from companies and workers' health care organizations who are currently active.
Sampling Method: Non-Probability Sample
Enrollment: 7300 (Estimated)
Dates: Start 2008-02; Primary Completion 2021-06 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
The influence of different factors on risk of sick leave for low back pain | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Mario Gestoso, MD, Principal Investigator — Kovacs Foundation,Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Guo HR, Tanaka S, Cameron LL, Seligman PJ, Behrens VJ, Ger J, Wild DK, Putz-Anderson V. Back pain among workers in the United States: national estimates and workers at high risk. Am J Ind Med. 1995 Nov;28(5):591-602. doi: 10.1002/ajim.4700280504. PMID 8561169
- [Background] Turner JA, Franklin G, Fulton-Kehoe D, Sheppard L, Wickizer TM, Wu R, Gluck JV, Egan K. Worker recovery expectations and fear-avoidance predict work disability in a population-based workers' compensation back pain sample. Spine (Phila Pa 1976). 2006 Mar 15;31(6):682-9. doi: 10.1097/01.brs.0000202762.88787.af. PMID 16540874
- [Background] Kovacs FM, Muriel A, Castillo Sanchez MD, Medina JM, Royuela A; Spanish Back Pain Research Network. Fear avoidance beliefs influence duration of sick leave in Spanish low back pain patients. Spine (Phila Pa 1976). 2007 Jul 15;32(16):1761-6. doi: 10.1097/BRS.0b013e3180b9f5f7. PMID 17632397
- [Derived] Seco-Calvo J, Royuela A, Rodriguez-Perez V, Kovacs F. Predicting low back pain-related absenteeism in the Spanish general working population. Occup Environ Med. 2026 Jan 21;82(11):547-555. doi: 10.1136/oemed-2025-110435. PMID 41443770